CLINICAL TRIAL: NCT00003842
Title: A Phase I Study of a Recombinant Chimeric Protein Composed of Circularly Permuted IL-4 and a Mutated Form of the Pseudomonas Exotoxin Termed IL-4(38-37)-PE38KDEL (IL-4 Toxin) for the Treatment of Recurrent Malignant Astrocytoma
Brief Title: IL-4(38-37)-PE38KDEL Immunotoxin in Treating Patients With Recurrent Malignant Astrocytoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Barrett Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067001; UCMC-981061; NBI-3001-9802; NCI-V99-1536
Record Dates: First submitted 1999-11-01; First posted 2004-09-14 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 1999-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — interleukin-4-Pseudomonas exotoxin; Surgical Procedures, Operative

INTERVENTIONS:
Biological: interleukin-4 PE38KDEL cytotoxin
Drug: isolated perfusion
Procedure: surgical procedure

SUMMARY:
RATIONALE: IL-4(38-37)-PE38KDEL immunotoxin may locate tumor cells and kill them without harming normal cells. This may be an effective treatment for recurrent malignant astrocytoma.

PURPOSE: Phase I trial to study the effectiveness of IL-4(38-37)-PE38KDEL immunotoxin in treating patients who have recurrent malignant astrocytoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of intratumorally infused IL-4(38-37)-PE38KDEL immunotoxin in patients with recurrent malignant astrocytoma. II. Determine the safety of this regimen in these patients. III. Determine preliminarily any efficacy of this regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study. Patients undergo a stereotactic biopsy under MR/CT guidance. Catheters are then placed into the tumor under stereotactic guidance. The catheter is filled with IL-4(38-37)-PE38KDEL immunotoxin (IL-4 toxin), with infusion beginning 24 hours after catheter insertion. The IL-4 toxin is infused over 4 days. The catheter is removed 45 minutes after the infusion is completed and a MR scan is performed. Cohorts of 3 patients each receive escalating doses of IL-4 toxin until the maximum tolerated dose (MTD) is reached. The MTD is defined as the dose preceding the dose at which 2 of 3 patients experience dose limiting toxicity. Patients are followed every 4 weeks for 16 weeks, then every 8 weeks for up to 3 years.

PROJECTED ACCRUAL: Approximately 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent glioblastoma or anaplastic astrocytoma Stereotactically accessible, enhancing mass no greater than 50 mL total volume by MRI No significant mass effect Recent craniotomy allowed No anaplastic oligodendroglioma No tumors of the brainstem, cerebellum, or both hemispheres No diffuse subependymal or CSF disease If on stable or increasing dose of steroid, must have evidence of increasing contrast enhancement by MRI or CT scan Prior external beam radiotherapy required

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9.5 g/dL Hepatic: Bilirubin less than 2 mg/dL AST and ALT less than 2 times upper limit of normal (ULN) PT/PTT no greater than ULN Renal: Creatinine less than 2 mg/dL Other: Not pregnant Negative pregnancy test Fertile patients must use effective contraception No systemic diseases to cause unacceptable anesthetic/operative risk No active infection requiring treatment No unexplained febrile illness

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent blood or platelet transfusions Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics Medically able to undergo surgery Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1999-03

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E. Warnick, MD, Study Chair — Barrett Cancer Center
Locations (10):
- United States (10):
  - University of Southern California, Healthcare Consultation Center, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Neuro-Oncology Service, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Laboratory of Molecular Biology, Bethesda, Maryland
  - Food and Drug Administration, Rockville, Maryland
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Charlotte Neurosurgical Associates, Charlotte, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio